CLINICAL TRIAL: NCT04937374
Title: Efficacy and Tolerability of Rehmannia Glutinosa Leaf Extract in the Treatment of Acne Vulgaris: a Double Blinded, Randomized, Placebo-controlled Clinical Trial
Brief Title: Efficacy and Tolerability of Rehmannia Glutinosa Leaf Extract in the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NS/201101/REHGLU/AV
Record Dates: First submitted 2021-05-31; First posted 2021-06-24 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Arm 1: Rehmannia Glutinosa leaf extract
  Arm 2: Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehmannia glutinosa leaf extract (Active Comparator): One capsule to be taken after breakfast for 56 days
  Interventions: Other: Rehmannia glutinosa leaf extract
- Microcrystalline Cellulose (MCC) (Placebo Comparator): One capsule to be taken after breakfast for 56 days
  Interventions: Other: Microcrystalline Cellulose (MCC)

INTERVENTIONS:
Other: Rehmannia glutinosa leaf extract — One capsule to be taken after breakfast.
  Arms: Rehmannia glutinosa leaf extract
Other: Microcrystalline Cellulose (MCC) — One capsule to be taken after breakfast.
  Arms: Microcrystalline Cellulose (MCC)

SUMMARY:
In this study, The Investigator will be assessing the efficacy and tolerability of Rehmannia glutinosa Libosch leaf-based extract formulation consumption on the treatment of Acne Vulgaris in a randomized, double-blind, placebo-controlled study for the duration of 56 days.

DETAILED DESCRIPTION:
In this study, The Investigator will be assessing the efficacy and tolerability of Rehmannia glutinosa Libosch leaf-based extract formulation consumption on the treatment of Acne Vulgaris in a randomized, double-blind, placebo-controlled study. The participants will consume one capsule per day containing active ingredient for the duration of 56 days. Throughout the duration of the clinical trial, The Investigator will be studying the formulation's effects on the change in the Global Acne Grading System (GAGS) score, facial sebum secretion, the number and irritability of inflammatory lesions, quality of life via the Acne-QoL questionnaire, skin wrinkle severity through the Modified Fitzpatrick Wrinkle Severity Scale (MFWS) and the percentage population of responders at the end of the study. The Investigator will also assess the change in skin radiance, luminosity, smoothness, texture, firmness, and skin hydration through a participant based self-assessment questionnaire as well as the safety and tolerability of the formulation through a global evaluation by the participants and the investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18 to 35 years
2. Body Mass Index (BMI) in the range of ≥ 18.5 to ≤ 29.9 kg/m2.
3. Moderate to severe acne as per GAGS (defined with a score of 19 to 38)
4. Participants ready to continue usual skin care regime till the entirety of study duration.
5. Participant willing to abstain Anti-acne preparations (creams, face wash, home remedies, etc) throughout the study.
6. Participants must be ready to abstain from any food supplements or medications and other related products apart from the ones allowed during the study period.
7. Participants must be willing to complete all study designated questionnaires and diaries or any other related procedures or requirements.
8. Participants having the ability to understand and sign a written informed consent form.

Exclusion Criteria:

1. Unwilling to forgo any aesthetic or dermatological treatments or procedures during the study period.
2. Consumption of any over-the-counter or prescribed oral anti-acne medications during the last 3 months prior to screening
3. Currently applying any over-the-counter or prescribed anti-acne medication including, but not limited to, retinoic acid or benzoyl peroxide over the past 3 months prior to screening.
4. Participants who have used facial, topical or injectable steroids 6 weeks prior to screening and during the study.
5. Females suffering from Polycystic Ovary Syndrome (PCOS).
6. Participant using oil and oil-based preparations for skin.
7. Consumptions of any herbal preparation, supplements, nutritional therapy or any other medications that is expected to improve acne over the past two weeks from randomization.
8. History of Hormonal imbalance
9. Abnormal Thyroid Stimulating Hormone (TSH) value which is < 0.35 or > 4.94 µIU/mL.
10. Participant with high caffeine consumption, (defined as >3 cups of coffee consumption in a day).
11. Topical or systemic use of antifungals and antibiotics in the previous 2 weeks prior to screening.
12. Participant having extremely oily food habits.
13. Participants taking drugs known to be photosensitizers including, but not limited to, phenothiazines, amiodarone, quinine, thiazides, tetracyclines, sulphonamides, quinolones
14. Known sensitivity to the investigational product or any excipients of the drug product.
15. Smoking or using any tobacco products.
16. Having a history of chronic skin allergies.
17. History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.
18. Participation in other clinical trials in last 30 days prior to screening
19. Participants with substance abuse problems (within 2 years) defined as:

    * Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
    * High-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week for women.
20. Patients who have clinically significant following severe illness (i.e., Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, gastrointestinal diseases, etc.)
21. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
22. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Acne severity: The global acne grading system | Day 0 Day 28 and Day 56
  Acne lesions will be counted separately for all the six locations. Then the acne score (S) will be multiplied with the area factor (F) to get local score of that particular area. All six local scores will be summed to get the total scores. The total acne severity scores will be obtained on day 0, day 28, and day 56. The change in acne severity of all the enrolled participants will be assessed after 28 and 56 days of supplementation from baseline (Day 0) and in comparison to placebo.

SECONDARY OUTCOMES:
Count of inflammatory acne lesions | Day 0 Day 28 and Day 56
  Acne vulgaris involves complications of pilosebaceous unit that causes inflammatory lesions (papules, pustules, and nodules).
  Inflammatory acne lesions are manifested by typical signs of inflammation i.e., swelling, redness, pain and heat.
  All the inflammatory acne lesions on the face will be counted on day 0, 28 and day 56.
  Any change in the number of these lesions on day 28 and 56 will be compared with baseline and placebo.
Sebum secretion | Day 0 Day 28 and Day 56
  Change in the facial sebum secretion will be assessed by Sebumeter® SM 815. decreased value interprets betterment of acne from Day 0 to Day 28 and Day 56 in comparison to Investigational product with placebo
Acne Quality of life questionnaire | Day 0 Day 28 and Day 56
  Acne-QoL consist of 19 items stratified in four subscales; Self-perception, Role-emotional, Role-social, and Acne symptoms.
  The QoL of such participants will be assessed using Acne-Specific Quality of Life Questionnaire (Acne-QoL) questionnaire.
  The total score varies from 0 to 114, distributed as follows: 0- 30 (self-perception), 0-24 (role-social), 0- 30 (role-emotional), and 0-30 (acne symptoms). A higher score reflects better health related QoL .
Percentage responders | Day 0 Day 28 and Day 56
  The participants' acne severity will be assessed using GAGS on day 0, 28 and 56. Participants will be declared as responders based on the improvement in acne severity as per GAGS severity grading system (based on total scores). Participants with improvement in acne severity by one grade or more as per GAGS on day 28 and 56 in comparison to baseline (Day 0) will be considered as responders. Percentage population of these responders will be evaluated in comparison to placebo
Pain VAS | Day 0 Day 28 and Day 56
  A VAS is an scale that measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is used regularly in clinical research studies for measuring the intensity or frequency of various symptoms. In the present study, a similar VAS will be used for assessment of physical symptoms associated with inflammatory acne lesions i.e., pain. The participant will be asked to mark the their severity of lesion pain as per the last 7 days on a 0 - 100 mm VAS scale on day 0, 28 and 56, where 0 - is no pain at all and 100 - is unbearable pain
Modified Fitzpatrick Wrinkle Severity Scale | Day 0 Day 28 and Day 56
  Changes in the wrinkle class from Class 3.0 indicated worst means Deep wrinkle. Deep and furrow wrinkle; more than 3-mm wrinkle depth to Class 0 indicates Good means No wrinkle. No visible wrinkle; continuous skin line.
Skin parameters using a participant based self-assessment questionnaire | Day 0 Day 28 and Day 56
  Highest Score represents Better and lowest Score represents Worst
Global evaluation of the efficacy by investigator | Day 56
  The investigator will assess on a scale of 0 (Very poor) to 4 (Excellent) as to how beneficial or vice-versa was the treatment experience over the study period on day 56. The outcomes will be evaluated in comparison to placebo
Itch VAS | Day 0 Day 28 and Day 56
  A VAS is an scale that measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is used regularly in clinical research studies for measuring the intensity or frequency of various symptoms. In the present study, a similar VAS will be used for assessment of physical symptoms associated with inflammatory acne lesions i.e., Itch. The participant will be asked to mark the their severity of lesion itch as per the last 7 days on a 0 - 100 mm VAS scale on day 0, 28 and 56 where 0 - is no itch at all and 100 - is unbearable itch.
Global evaluation of the tolerability by Participant | Day 56
  The Participant will self-assess on a scale of 0 (Very poor) to 4 (Excellent) as to how beneficial or vice-versa was the treatment experience over the study period on day 56. The outcomes will be evaluated in comparison to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Manjiri Jagtap, M.B.B.S, D.N.B, Principal Investigator — SKIN CURE N CARE
Locations (1):
- Skin cure and care clinic, Thane, Maharashtra, India